CLINICAL TRIAL: NCT06556446
Title: Safety and Efficacy of Intravenous Thrombolysis in Patients With Ischemic Stroke and Recent Ingestion of Direct Oral Anticoagulants: the DOAC - International Thrombolysis (DO-IT) Cohort Study
Brief Title: Intravenous Thrombolysis in Patients With Ischemic Stroke and Recent Ingestion of Direct Oral Anticoagulants
Acronym: DO-IT Cohort
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Stroke Trialist Association (Unknown); Swiss Stroke Registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-01175
Record Dates: First submitted 2024-06-24; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Ischemic Stroke
Keywords: DOAC (Direct Oral AntiCoagulants); NOAC (Novel Oral AntiCoagulants); Anticoagulation; r-tPA (tissue-type plasminogen activator); Alteplase; Tenecteplase; Rivaroxaban; Apixaban; Dabigatran; Edoxaban
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- DOAC+IVT: Acute ischemic Stroke patients with recent DOACs intake receive IVT.
  Interventions: Drug: Tenecteplase and Alteplase
- DOAC: Acute ischemic Stroke patients with recent DOAC intake do not receive IVT.
- IVT Controls: Acute ischemic Stroke patients without recent DOAC intake receive IVT.

INTERVENTIONS:
Drug: Tenecteplase and Alteplase — The timepoints, dose, and type of IVT will be collected as well as any complications occuring.
  Groups: DOAC+IVT

SUMMARY:
DO-IT is an international, prospective observational registry evaluating whether the administration of intravenous thrombolysis (IVT) is safe and improves functional outcome in ischemic stroke patients with recent direct oral anticoagulant (DOAC) intake. For this purpose, information on 2800 adult participants experiencing an acute ischemic stroke will be obtained at several high-volume international stroke centers and divided into three groups: IVT with recent DOACs intake (DOAC+IVT), and recent DOAC intake not receiving IVT (DOAC) as well as anonymized patients without DOAC receiving IVT. The patients are followed up for 90 days after the index event. treatment recommendations from the described observations. The investigators hypothesize that also more liberal decisions for IVT in patients with recent DOAC intake are not associated with an increased risk for symptomatic intracerebral hemorrhage (sICH) and result in better functional outcome at 3 month.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of acute ischemic stroke with indication for IVT according to applicable guidelines
2. Time from symptom onset or last known well <12 hours
3. Admission NIHSS of 2 points or more
4. either DOAC ingestion within 48 hours prior to expected timepoint of IVT bolus, or patient with an ongoing prescription of DOAC, but exact timepoint of last intake not verifiable in the emergency setting. (regardless of whether intravenous thrombolysis was given) OR DOAC prescription (any intake within the last 7 days) and receiving intravenous thrombolysis
5. Informed consent (if obtainable and in those international sites where this is legally required) for the prospective part

Exclusion Criteria:

1. Patient refused the use of biological data for research purposes (Switzerland)
2. Any acute or subacute intracranial hemorrhage (ICH) identified by admission CT or MRI on brain scan
3. Documentation of any other absolute contraindications to IVT in the medical record
4. Significant pre-stroke disability (mRS score of 5), including known advanced dementia
5. Known (serious) sensitivity to Alteplase/Tenecteplase or any of the excipients
6. Pregnancy or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The in- and exclusion criteria emulate a target trial, thus the investigators want to study a population that is - except from recent DOAC ingestion - eligible for IVT as per standard of care.
Sampling Method: Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with symptomatic intracerebral hemorrhage (sICH) | Within 36 hours after IVT
  Defined as worsening of at least 4 points on the National Institutes of Health Stroke Scale and attributed to radiologically evident intracranial hemorrhage.
Dichotomized good functional outcome (mRS 0-2) | At day 90 or return to baseline (+/- 2 weeks) after admission
  Modified Rankin Scale from 0 (no disability) to 6 (death)

SECONDARY OUTCOMES:
Rate of IVT among IVT-eligible DOAC patients | Through study completion, an average of 2 years
  To determine the rate of IVT in eligible patients with acute ischemic stroke and recent DOAC intake.
All-cause mortality, major bleeding and orolingual edema | From date of randomization until the date of all-cause mortality, major bleeding or orolingual edema, whichever came first, assessed up to 7 days.
Categorical shift in the modified Rankin Scale (mRS) | At Day 90 (+/-2 weeks) after admission
  Modified Rankin Scale from 0 (no disability) to 6 (death)
Stroke severity (NIHSS) | At 24 hours ±8 hours
  National Institutes of Health Stroke Scale from 0 (no symptoms) to 39 (most severe symptoms)
Ischemic stroke volume at 24 hours (mL) | At 24 hours ±8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meinel, MD, PhD, Study Director — Insel Gruppe AG, University Hospital Bern
Locations (33):
- Medical University of Innsbruck, Innsbruck, Austria
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Leuven, Leuven
- The University of British Columbia | Vancouver General Hospital, Vancouver, Canada
- CHU Caen, Caen, France
- Germany (2):
  - Nordwest-Krankenhaus Sanderbusch, Sanderbusch
  - Universitäsklinikum Tübingen, Tübingen
- Dept. of Medicine, University of Thessaly, Larissa, Thessaly, Greece
- Italy (4):
  - A.O.R.N. Antonio Cardarelli Hospital, Naples
  - Ospedali Riuniti Hospital, Palermo
  - Ospedale "Bufalini", Cesena, Perugia
  - AUSL-IRCCS di Reggio Emilia, Reggio Emilia
- Akershus Hospital, Oslo, Norway
- Hospital de Egas Moniz, Lisbon, Portugal
- Clinical Centre of Serbia, University Hospital Belgrade, Belgrade, Serbia
- National University Hospital, Singapore, Singapore
- Ljubljana University Medical Centre, Ljubljana, Slovenia
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
- Switzerland (12):
  - Kantonsspital Aarau, Aarau
  - Unispital Basel, Basel
  - Inselspital Bern, University Hospital Bern, Bern
  - HFR Fribourg, Fribourg
  - University Hospital Geneva, Geneva
  - CHUV Lausanne, Lausanne
  - Kantonsspital Lucerne, Lucerne
  - EOC Lugano, Lugano
  - Hôpital Neuchâtelois, Neuchâtel
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hirslanden Zurich, Zurich
  - University Hospital Zurich, Zurich
- United Kingdom (2):
  - Imperial College London NHS Trust, London
  - King'S College Hospital Nhs Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
IPDMA of similar observational cohort studies is planned.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of primary study results
Access Criteria: Ethics clearance, agreement with the DO-IT collaboration about terms of use and authorship